CLINICAL TRIAL: NCT04024098
Title: An Epidemiological Survey of Cancer-related Fatigue Among Taiwanese Gynecologic
Brief Title: An Epidemiological Survey of Cancer-related Fatigue Among Taiwanese Gynecologic Cancer Patients
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, CHING-CHOU TSAI, Attending physician, Chang Gung Memorial Hospital
Other Study IDs: CRF-CGMH01
Record Dates: First submitted 2019-07-08; First posted 2019-07-18 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Fatigue
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aim is to examine the prevalence, severity, and management of CRF among Taiwanese gynecologic cancer patients.

DETAILED DESCRIPTION:
The cross-sectional survey is conducted at oncology inpatients unit and outpatients clinics of hospitals in Taiwan. Furthermore, the results will elucidate not only the epidemiology of CRF in Taiwan, but will supply physicians with more understanding about CRF, and help them to enhance the quality on cancer care to being perfected in the future.

ELIGIBILITY:
Inclusion Criteria:

* Patients who signed the informed consent form
* The age of eligible patients should be ≥ 20 years old.
* Inpatients or outpatients who have been given a diagnosis of gynecologic cancer.
* Able to communicate verbally and completely fill out the questionnaires

Exclusion Criteria:

* Patients who have been given a diagnosis of cognitive impairment are unable to complete the questionnaires

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: gynecologic cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-07-11 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Cancer-related fatigue evaluation-1 | 10 minuts
  ICD-10 Fatigue Criteria
Cancer-related fatigue evaluation-2 | 8 minuts
  Brief Fatigue Inventory-Taiwan Form (BFI-T)
Symptoms and Quality of Life Assessments-1 | 4 minuts
  Functional Assessment of Cancer Therapy-General quality of life questionnaire (FACT-G7)
Symptoms and Quality of Life Assessments-2 | 5 minuts
  cancer symptom survey (self-designed questionnaire)

CONTACTS AND LOCATIONS:
Overall Officials: CHING-CHOU TSAI, Dr., Principal Investigator — Kaohsiung Chan Gung Memorial Hospital
Locations (1):
- Kaohsiung Chan Gung Memorial Hospital, Kaohsiung City, Taiwan